CLINICAL TRIAL: NCT01192737
Title: Cohort Study to Evaluate Clinical Expression and Maternofetal Consequences of A/H1N1 Influenza in Pregnant Women
Brief Title: "COhort Study on A/H1N1 FLU During PREGnancy"
Acronym: COFLUPREG
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C09-24; 2009-015160-34 (EudraCT Number)
Record Dates: First submitted 2010-07-20; First posted 2010-09-01 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2012-04

CONDITIONS: Influenza; Pregnancy
Keywords: pandemic; A/H1N1; pregnancy; cohort; vaccine; Influenza and Pregnancy
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, cord blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to measure the incidence of A/H1N1 Influenza infection in the mother and her child and to identify the determinants in pregnant women during pandemic period in three public maternities in Paris, France.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Pregnancy between 12 and 35 weeks of gestation, going in one of the following maternity cares: Port Royal, Necker, Saint Vincent de Paul
* Provides written informed consent
* Speaks and understands French
* Covered by French Social Security

Exclusion Criteria:

* Not covered by French Social Security
* Previous H1N1 influenza (virologically documented)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 919 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Frequency of A/H1N1 Influenza virus infection in pregnant women and impact of Flu on pregnancy outcome. | 1 year

SECONDARY OUTCOMES:
Safety of Flu vaccine | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, PhD, Principal Investigator — CIC de Vaccinologie Cochin Pasteur
Locations (3):
- France (3):
  - Maternité Necker-Brune, Paris
  - Maternité Port Royal, Paris
  - Maternité Saint Vincent de Paul, Paris

REFERENCES:
- [Result] Launay O, Krivine A, Charlier C, Truster V, Tsatsaris V, Lepercq J, Ville Y, Avenell C, Andrieu T, Rozenberg F, Artiguebielle F, Treluyer JM, Goffinet F; Inserm COFLUPREG Study Group. Low rate of pandemic A/H1N1 2009 influenza infection and lack of severe complication of vaccination in pregnant women: a prospective cohort study. PLoS One. 2012;7(12):e52303. doi: 10.1371/journal.pone.0052303. Epub 2012 Dec 27. PMID 23300637